CLINICAL TRIAL: NCT02229903
Title: A Prospective Double Blind Randomized Controlled Trial to Evaluate the Safety and Efficacy of the Deep Transcranial Magnetic Stimulation (dTMS) in Obsessive-Compulsive Subjects
Brief Title: An Evaluation of the Safety and Efficacy of the dTMS Treatment for OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP-OCD-01
Record Dates: First submitted 2014-08-07; First posted 2014-09-03 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2017-02

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active DTMS Treatment (Active Comparator): Active DTMS Treatment constitutes the Deep Transcranial Magnetci Stimulation (DTMS) which is a new form of TMS which allows direct stimulation of deeper neruonal pathways than the standard TMS. The DTMS coil is designed to allow deeper brain stimulation without significant increase of electric fields included in superficial cortical regions.
  Interventions: Device: Active DTMS Treatment
- Sham Treatment (Sham Comparator): The Sham Treatment consists of an electrical field which cannot invoke any action potentials and if no action potentials are induced, then the electric field is insignificant and there is no treatment effect on the brain.
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Active DTMS Treatment — H-coil Deep TMS 29 TMS treatments over 6 weeks.
  Arms: Active DTMS Treatment
Device: Sham Treatment — 29 treatments over 6 weeks.
  Other Names: Deep TMS Sham treatment
  Arms: Sham Treatment

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the Deep TMS (DTMS) treatment in subjects with OCD. The device technology is based on the application of deep brain TMS by means of repetitive pulse trains at a predetermined frequency. The Brainsway DTMS study is a randomized, 10 week, double blind, multi-center trial comparing active DTMS treatment to sham treatment.

DETAILED DESCRIPTION:
The OCD study will compare one group of OCD subjects receiving DTMS treatment (HAC-coil) to a second group of OCD subjects receiving sham treatment (sham coil). The treatment group will receive 5 weeks of daily DTMS treatments followed by 4 treatments in week 6, for a total of 29 treatment sessions. The control group will receive the same treatments with a sham coil. Subjects may continue to take SSRI medications (if prescribed) and any other antidepressant medications will be tapered down prior to the first treatment. SSRI medications approved for OCD include Fluoxetine (Prozac, Sarafem, Symbyax), Fluvoxamine (Luvox, Luvox CR), Paroxetine (Paxil, Paxil CR, Pexeva) and Sertraline (Zoloft). Efficacy will be assessed using the Yale-Brown Obsessive Compulsive Scale score (YBOCS), as well as other efficacy scales. Safety will be assessed by monitoring of adverse events, vital signs, physical and neurological examination and using certain safety questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- • Outpatients

* Men and women 22-68 years of age.
* Subjects diagnosed as suffering from OCD according to the DSM-IV-TR.
* Subjects with at least moderate OCD, rating a YBOCS score of >20.
* Subjects are maintained on SSRI medication at at least a therapeutic dosage for at least 2 months prior to study entry and for the duration of the trial and/or subjects are maintained on psychotherapeutic behavioral intervention therapy (subjects undergoing CBT treatment must be in the maintenance stage (i.e., not during the assessment or skills acquisition or training stages).
* Subjects with negative responses on the Transcranial Magnetic Stimulation Safety Screening questionnaire (TASS).
* According to the treating physician the subject is compliant with taking medication, if applicable.
* Subject is capable and willing to provide informed consent.
* Subject is able to adhere to the treatment schedule.

Exclusion Criteria:

- • Subjects diagnosed according to the SCID I as suffering from any other Axis I diagnosis as the primary diagnosis.

* Subjects diagnosed according to the SCID II as suffering from severe Personality Disorder (excluding Obsessive Compulsive Personality Disorder) or hospitalized due to exacerbation related to borderline personality disorder.
* Present suicidal risk as assessed by the investigator using the Scale for Suicide Ideation (SSI), brief mental status exam and psychiatric interview or significant suicide risk based on HDRS-21 item 3 score of 3 or 4 or a history of attempted suicide in the past year.
* Subject has a history of epilepsy or seizure (EXCEPT those therapeutically induced by ECT) or history of such in first degree relatives.
* Subject has an increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes.
* Subject has a history of head injury necessitating cranial surgery or prolonged coma.
* Subject has a history of any metal in the head including the eyes and ears (outside the mouth).
* Subject has known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* Subject has a history of significant hearing loss.
* Subjects with significant neurological disorder or insult including, but not limited to:
* Any condition likely to be associated with increased intracranial pressure
* Subject has a history of substance abuse including alcoholism within the past 6 months (except nicotine and caffeine).
* Inadequate communication with the patient.
* Subject is currently participating in another clinical study or enrolled in another clinical study within 30 days prior to this study.
* Subjects who suffer from an unstable physical, systemic and metabolic disorder such as unstabilized blood pressure or acute, unstable cardiac disease.
* Subject is currently on any antidepressant medication other than SSRIs.
* Subject is currently on Clomipramine
* Subject has had previous treatment with TMS
* Women who are breast-feeding
* Women who are pregnant or with suspected pregnancy
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) score | 6 Weeks
  The primary objective of the study is to compare the change in Yale Brown Obsessive Compulsive Scale (YBOCS) scores from baseline to the 6 week (post-randomization) visit, between the two treatments groups.

SECONDARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS), Sheehan Disability Scale (SDS), Clinical Global Impression - Severity Scale (CGI-S), Clinical Global Impression - Improvement Scale (CGI-I) | 6 Weeks and 10 weeks
  The secondary effectiveness objectives of the study are:
  i. Change from baseline to 6 weeks in Yale Brown Obsessive Compulsive Scale (YBOCS) (and other assessment scale) scores, between treatment groups.
  ii. Response rate at 6 weeks in Yale Brown Obsessive Compulsive Scale (YBOCS) score from baseline, between treatment groups; iii.Partial Response rate at 6 weeks in Yale Brown Obsessive Compulsive Scale (YBOCS) score, between treatment groups; iv. Change from baseline to 10 weeks in above scales. v. Remission rates at 6 weeks between treatment groups.

OTHER OUTCOMES:
Number of adverse events, changes in vitals signs, physical and neurological results, changes in suicide scale and changes in cognitive scales | 10 Weeks
  Safety of the DTMS treatment as defined by maintained subject baseline, pre-treatment, physical and neurological examinations and lack of significant increase in suicide ideation measured by:
  * Vital signs
  * Physical and neurological examination
  * Scale for Suicide Ideation
  * Cognitive evaluation using the Mini-Mental State Exam (MMSE), Buschke Selective Reminding Test (BSRT) and Autobiographical Memory Interview - Short Form (AMI-S) scales
  * Any other adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, Prof, Principal Investigator — Tel Hashomer Hospital; Abraham Zangen, Prof, Principal Investigator — Soroka University Medical Center
Locations (12):
- United States (10):
  - University of California (UCLA), Los Angeles, California
  - University of California, San Diego, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - University of Chicago, Chicago, Illinois
  - Neuropharmacology Services, New York, New York
  - Mount Sinai Hospital, New York, New York
  - TMS Hope Center of Long Island, New York, New York
  - Lindner Center of HOPE, University of Cincinnati College of Medicine, Mason, Ohio
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada
- Tel Hashomer Hospital, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Harmelech T, Tendler A, Roth Y, Zangen A. Do comorbid OCD-MDD patients need two separate dTMS protocols? Brain Stimul. 2020 Jul-Aug;13(4):1000-1001. doi: 10.1016/j.brs.2020.03.014. Epub 2020 Mar 31. No abstract available. PMID 32380442
- [Derived] Crowell AL, Riva-Posse P, Holtzheimer PE, Garlow SJ, Kelley ME, Gross RE, Denison L, Quinn S, Mayberg HS. Long-Term Outcomes of Subcallosal Cingulate Deep Brain Stimulation for Treatment-Resistant Depression. Am J Psychiatry. 2019 Nov 1;176(11):949-956. doi: 10.1176/appi.ajp.2019.18121427. Epub 2019 Oct 4. PMID 31581800
- [Derived] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199